CLINICAL TRIAL: NCT05916534
Title: Brooklyn Digital Community Care Intervention to Address Unmet Social Needs and Optimize Engagement in Maternal Health Care
Brief Title: We Care About Brooklyn - A Digital Behavioral Intervention to Optimize Engagement in Maternal Healthcare
Acronym: WeCAB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: State University of New York - Downstate Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1R21NR020706-01 (NIH)
Record Dates: First submitted 2023-06-14; First posted 2023-06-23 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Maternal Health; Pregnant Women
Keywords: Digital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WeCAB Intervention (Experimental)
  Interventions: Behavioral: WeCAB Intervention
- Usual Care (No Intervention)

INTERVENTIONS:
Behavioral: WeCAB Intervention — The WeCAB intervention will use a dedicated WeCAB community health worker who will administer a social determinants of health (SDOH) tool and use digital care navigation to monitor closed loop referrals.
  Arms: WeCAB Intervention

SUMMARY:
The goal of this clinical trial is to test a behavioral intervention in pregnant women who identify as Black and live in Central Brooklyn. The main question it aims to answer is whether the WeCAB intervention leads to a net improvement in utilization of postpartum care compared to those receiving usual care.

The WeCAB group will have a dedicated WeCAB community health worker who will be trained in digital care navigation.

Researchers will compare the WeCAB group versus the group receiving usual care to see if the patients randomized to WeCAB will have higher rates of early post-partum care compared to patients in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants for the pilot RCT will be patients
* aged 18-49 years (childbearing age)
* residing in a Central Brooklyn zip code
* self-reporting as Black,
* who speak English or Haitian Creole, and
* plan to deliver or present for delivery at University Hospital at Downstate (UHD).
* In NYC, SMM increases incrementally with later entry into prenatal care (1st trimester: 208/10,000 deliveries; 2nd trimester: 252/10,000; 3rd trimester: 297/10,000; None: 575/10,000). 3 Accordingly, in order to capture the full range of SMM risk profiles for our pilot study, any pregnant patient/client visiting our clinics will be eligible for enrollment from 13 weeks gestation through delivery, thus allowing follow-up to 3 months post-partum within the 2-year study timeline.

Exclusion Criteria:

* Patients planning to move outside of New York City in the ensuing 3 months post-partum
* Patients demonstrating an impairment that limits their ability to provide informed consent.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-11-20 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Initiation of postpartum care | 13 weeks until 3 months postpartum
  Initiation of postpartum care within 6 weeks of delivery

SECONDARY OUTCOMES:
Maternal death | 13 weeks until 3 weeks postpartum
  Death of a woman while pregnant or within 42 days of termination of pregnancy, irrespective of the duration and site of the pregnancy, from any cause related to or aggravated by the pregnancy or its management but not from accidental or incidental causes.

CONTACTS AND LOCATIONS:
Overall Officials: Aimee Afable, PHD, Principal Investigator — SUNY Downstate
Locations (1):
- University Hospital at Downstate, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No